CLINICAL TRIAL: NCT04286971
Title: Preoperative Continuous Sciatic Perineural Analgesia, as a Bridge Therapy for Ischemic Pain, in Patients Undergoing Lower Limb Revascularization: a Retrospective Descriptive Study
Brief Title: Preoperative Continuous Sciatic Perineural Analgesia in Patients Undergoing Lower Limb Revascularization
Status: Completed | Type: Observational
Sponsor: Hospital Municipal Miguel Couto (Other)
Responsible Party: Principal Investigator, Rafael Mercante Linhares, Head of Anesthesiology and Pain Medicine Department, Hospital Municipal Miguel Couto
Other Study IDs: 25206319.3.0000.5279
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Ischemic Leg; Peripheral Vascular Disease
Keywords: continuous peripheral block; sciatic block; ischemic pain
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the pain score numerical rating, after sciatic analgesic continuous block, in patients with ischemic pain before surgery of limb revascularization. All patients received those blocks to control ischemic severe pain.

DETAILED DESCRIPTION:
Peripheral Obstructive Arterial Disease (PAD) is a disease with a prevalence of 10 to 25% in the population over 55 years, increasing with age, and may have disabling pain as a symptom, and sometimes the surgical approach is required. In the context of public hospital in Rio de Janeiro, where patients need to wait for surgery, the Anesthesiology and Acute Pain service routinely has sciatic nerve analgesic block in the popliteal region as a preoperative procedure.

The primary objective of the present study is to describe a series of cases where the technique was applied in order to relieve the pain of these patients, following the Pain Score Numerical rating as a reference. Secondary objectives will be to describe difficulties associated with the technique and possible associated adverse factors.

ELIGIBILITY:
Inclusion Criteria:

* preoperative continuous sciatic-popliteal nerve block
* lower limb angioplasty
* peripheral arterial disease;
* between 2017 and 2018 years;
* correct filling of numerical rating pain evaluation in the medical record

Exclusion Criteria:

* peripheral block to treat another pathology or condition in te same patient;
* peripheral block at another concomitant site (other than the popliteal);
* No adequate record of the care received in the medical record
* if medical record is not available during the data collection period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with lower limb isquemic pain caused by peripheral arterial disease in the preoperative period.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
change in numerical pain scale | 24 hours after placement of sciatic catheter
  Numerical Pain Scale (END) self-assessed by the patient before and after 24 hours of continuous analgesic block of the sciatic nerve, with infusion of levobupivacaine 0,125% or ropivacaine 0,2%. The scale score is 0-10 (0= no pain; 10 = pain as bad as can be)

SECONDARY OUTCOMES:
change in numerical pain scale | 72 hours after placement of sciatic catheter
  Numerical Pain Scale (END) self-assessed by the patient before and after 72 hours of continuous analgesic block of the sciatic nerve, with infusion of levobupivacaine 0,125% or ropivacaine 0,2%. The scale score is 0-10 (0= no pain; 10 = pain as bad as can be)
classification of technique difficulties | 72 hours after placement of sciatic catheter
  To report, qualitatively, the presence of variations or difficulties in the use of the technique, such as: failure of the technique (FT); existence of concomitant venous analgesia (VA); inadequate registration of the technique (IR)
classifications of possible complications | 72 hours after placement of sciatic catheter
  Report, qualitatively, the presence of possible complications, such as: hyperemia of the catheter insertion site (HC); the presence of pus (PUS); catheter displacement (CD)

CONTACTS AND LOCATIONS:
Locations (1):
- Rafael M Linhares, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luiten WE, Schepers T, Luitse JS, Goslings JC, Hermanides J, Stevens MF, Hollmann MW, van Samkar G. Comparison of continuous nerve block versus patient-controlled analgesia for postoperative pain and outcome after talar and calcaneal fractures. Foot Ankle Int. 2014 Nov;35(11):1116-21. doi: 10.1177/1071100714546640. Epub 2014 Aug 12. PMID 25116132
- [Background] Thomas K, Barrett B, Tupper R, Dacenko-Grawe L, Holm K. Pain management after total knee arthroplasty: a case-control study of continuous nerve block therapy. Orthop Nurs. 2014 Sep-Oct;33(5):268-76. doi: 10.1097/NOR.0b013e3182879bd9. PMID 25362748
- [Background] Gelfand HJ, Ouanes JP, Lesley MR, Ko PS, Murphy JD, Sumida SM, Isaac GR, Kumar K, Wu CL. Analgesic efficacy of ultrasound-guided regional anesthesia: a meta-analysis. J Clin Anesth. 2011 Mar;23(2):90-6. doi: 10.1016/j.jclinane.2010.12.005. PMID 21377070
- [Background] Compere V, Cornet C, Fourdrinier V, Maitre AM, Duparc F, Biga N, Dureuil B. [Evaluation of continuous nerve block for postoperative pain management in orthopaedic surgery]. Ann Fr Anesth Reanim. 2005 Jul;24(7):795-801. doi: 10.1016/j.annfar.2005.04.025. French. PMID 15949910
- [Background] Aubuchon A, Arnold WD, Bracewell A, Hoyle JC. Sciatic neuropathy due to popliteal fossa nerve block. Muscle Nerve. 2017 Oct;56(4):822-824. doi: 10.1002/mus.25622. Epub 2017 Jun 6. PMID 28214338
- [Background] Dingemans SA, de Ruiter KJ, Birnie MFN, Goslings JC, van Samkar G, Schepers T. Comparable Postoperative Pain Levels Using 2 Different Nerve Blocks in the Operative Treatment of Displaced Intra-articular Calcaneal Fractures. Foot Ankle Int. 2017 Dec;38(12):1352-1356. doi: 10.1177/1071100717730337. Epub 2017 Sep 16. PMID 28918661
- [Background] Kim NY, Lee KY, Bai SJ, Hong JH, Lee J, Park JM, Kim SH. Comparison of the effects of remifentanil-based general anesthesia and popliteal nerve block on postoperative pain and hemodynamic stability in diabetic patients undergoing distal foot amputation: A retrospective observational study. Medicine (Baltimore). 2016 Jul;95(29):e4302. doi: 10.1097/MD.0000000000004302. PMID 27442676
- [Background] Dao T, Amaro-Driedger D, Mehta J. Successful treatment of Raynaud's syndrome in a lupus patient with continuous bilateral popliteal sciatic nerve blocks: a case report. Local Reg Anesth. 2016 Jun 15;9:35-7. doi: 10.2147/LRA.S97111. eCollection 2016. PMID 27366104
- [Result] Joshi G, Gandhi K, Shah N, Gadsden J, Corman SL. Peripheral nerve blocks in the management of postoperative pain: challenges and opportunities. J Clin Anesth. 2016 Dec;35:524-529. doi: 10.1016/j.jclinane.2016.08.041. Epub 2016 Oct 20. PMID 27871587